CLINICAL TRIAL: NCT04289142
Title: Cognitive Outcomes After Dexmedetomidine Sedation in Cardiac Surgery Patients: CODEX Trial
Brief Title: Cognitive Outcomes After Dexmedetomidine Sedation in Cardiac Surgery Patients
Acronym: CODEX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: London Health Sciences Centre (Other); University Health Network, Toronto (Other); McMaster University (Other); Canadian Institutes of Health Research (CIHR) (Other Government); The Dana Foundation (Other); Brain Canada (Other); Alzheimer's Association (Other); Hamilton Health Sciences Corporation (Other); University of Saskatchewan (Other); Fraser Health (Other); Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1743
Record Dates: First submitted 2019-10-09; First posted 2020-02-28 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-07

CONDITIONS: Delirium; Cognitive Dysfunction; Cognition Disorder; Neurocognitive Disorders; Mental Disorders; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms; Dexmedetomidine; Hypnotics and Sedatives; Central Nervous System Depressants; Physiological Effects of Drugs; Analgesics, Non-Narcotic; Analgesics; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Delirium; Cognitive Dysfunction; Cognition Disorders; Neurocognitive Disorders; Mental Disorders; Confusion; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Signs and Symptoms | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Hydrochloride Group (Active Comparator): Patients will receive a loading dose of 1.2 μg/kg dexmedetomidine prior to transfer to CVICU over 20-60 min immediately postoperative, followed by continuous infusion of 0.3 μg/kg/h for up to 12 hours or until patient is ready for discharge from CVICU (whichever is earlier). Any additional sedatives necessary at the discretion of ICU.
  Interventions: Drug: Dexmedetomidine Hydrochloride Group
- Standard of Care Group (No Intervention): Standard sedation protocols will be followed at the discretion of the attending physician.

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride Group — Dexmedetomidine will be initiated prior to transfer to the CVICU with loading dose of 1.2 ug/kg over approximately 20-60 minutes. This will be followed by an infusion at 0.3 ug/kg/h in CVICU for up to 12 hours from the time DEX infusion started or until the patient is ready for discharge from the CVICU (whichever is earlier). Any additional sedatives necessary at the discretion of ICU.
  Other Names: Dexmedetomidine Hydrochloride
  Arms: Dexmedetomidine Hydrochloride Group

SUMMARY:
Anesthesia is a drug induced, reversible, comatose state that facilitates surgery and it is widely assumed that cognition returns to baseline after anesthetics have been eliminated. However, many patients have persistent memory impairment for weeks to months after surgery. Cardiac surgery appears to carry the highest risk of postoperative cognitive dysfunction (POCD). These cognitive deficits are associated with increased mortality, prolonged hospital stay and loss of independence. The investigators propose to investigate the role of Dexmedetomidine (DEX) in preventing long-term POCD after cardiac surgery and enhancing early postoperative recovery. It is anticipated that DEX will be the first effective preventative therapy for POCD, improve patient outcomes, and reduce length of stay and healthcare costs.

DETAILED DESCRIPTION:
Dexmedetomidine (DEX), a highly potent and selective α2-adrenoceptors (α2R) agonist used in clinical practice for sedation, analgesia, and anxiolysis, was recently shown to have beneficial effects on early cognitive changes by reducing delirium in humans. It also reduced memory impairment after surgery and isoflurane anesthesia, both in elderly mice (20-22 months) and in pups exposed to anesthesia in the early postnatal period. Importantly, co-treatment with DEX has been shown to restore learning and memory function in rats exposed to propofol in utero. Therefore, the investigators set out to investigate whether DEX has an effect on cognitive dysfunction months after surgery and whether it accelerates cognitive recovery from anesthesia and surgery.

This is a double blinded, multi-site trial facilitated by Clinical Trials Ontario (CTO). Participants will be randomized 1:1 in permuted blocks of 4 to 8. The randomization sequence will be computer generated and stratified by 2 factors, planned procedure (CABG/CABG + valve or valve only procedure) and study site.

In hospital outcomes include delirium (assessed twice daily post-operative day (POD) 0-10, death, hemodynamic instability requiring vasopressors, time to extubation, re-intubation (and reason), length of stay (in Cardiovascular Intensive Care Unit and total hospital), POCD, depressive symptoms between POD 4-10, post-operative complications (infection [surgical site, sepsis, pneumonia], myocardial infarction, renal replacement therapy, re-operation, cumulative opioid consumption (to POD 5), in-hospital mortality.

Post-operative outcomes include POCD (3/6/12 months), depression (3/6/12 months), mild cognitive impairment (MCI) at 3/6/12 months (defined as 1-2 standard deviations below age matched controls), persistent surgical site pain at sternotomy/thoracotomy/graft harvest site (Brief Pain Inventory, 3/6/12 months), recovery (3,6, 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Planned CABG (+/- valve, including off-pump) or valve replacement via sternotomy/thoracotomy, with initial recovery in the Cardiovascular Intensive Care Unit (CVICU)
* Age ≥60

Exclusion Criteria:

* Lack of patient consent
* Pre-operative major cognitive dysfunction (CogState Brief Battery score < 80) at screening
* Aortic arch replacement/re-implantation (surgery requiring hypothermic circulatory arrest, e.g. Bentall procedure)
* Allergy/contraindication to dexmedetomidine (untreated 2nd degree type 2 or 3rd degree heart block (pacemaker), cirrhosis, HR < 50 , grade 4 LV, renal failure or on renal replacement therapy)
* Unlikely to comply with study assessments (e.g. no fixed address, cannot complete cognitive tests at the 3, 6, and 12 month time points)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative cognitive dysfunction | 3 months
  Presence of POCD assessed by CogState Brief Battery (CBB)

SECONDARY OUTCOMES:
Post-operative cognitive dysfunction (POCD) at 1 week, 6 months, 12 months after surgery | 1 week, 6 and 12 months
  POCD assessed by CogState Brief Battery (CBB)
Delirium | Anytime up to post-operative day 10
  Confusion Assessment Method (CAM/CAM-ICU) or Intensive Care Delirium Screening Checklist (ICDSC), binary scale to determine if delirium is present or absent
Length of stay | An average of 5 -14 days
  ICU and total hospital stay
Depressive symptoms | 3, 6, and 12 months
  Evaluated by PHQ-9 (Patient Health Questionnaire, scale 0-27, higher score is worse outcome)
Persistent Surgical Site Pain | 3, 6, and 12 months
  Evaluated by Brief Pain Inventory
Quality of Surgical Recovery | 3, 6, 12 months
  Evaluated by QoR- (Quality of Recovery) 40 questionnaire (scale: 0-200, higher is better outcome)
Mild Cognitive Impairment | 3, 6, and 12 months
  Presence of MCI assessed by CogState Brief Battery (CBB)
In-hospital mortality for index surgery | through initial inpatient admission, average of 1 week
  death before hospital discharge after surgery
Opioid consumption to POD 4 | 4 days
  Cumulative opioid consumption
Time to extubation | through ICU stay, average of 12 hours
  Time from ICU arrival to cessation of mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Choi, MD,MSc,FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (8):
- Canada (8):
  - Royal Columbian Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - London Health Sciences, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Laval University, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
All de-identified participants data collected during this trial that underlie the results reported in the publication(s) will be available upon request after publication of the primary results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available upon request immediately after publication of the primary results. No end date.
Access Criteria: Direct request to PI. Anyone who wishes to access the data.

REFERENCES:
- [Derived] Choi S, Jerath A, Jones P, Avramescu S, Djaiani G, Syed S, Saha T, Kaustov L, Kiss A, D'Aragon F, Hedlin P, Rajamohan R, Couture EJ, Singh A, Mapplebeck JC, Wong S, Orser BA. Cognitive Outcomes after DEXmedetomidine sedation in cardiac surgery: CODEX randomised controlled trial protocol. BMJ Open. 2021 Apr 13;11(4):e046851. doi: 10.1136/bmjopen-2020-046851. PMID 33849856